CLINICAL TRIAL: NCT00754520
Title: A Multi-center Prospective Randomized Control Trial to Compare Two Articulating Bearing Surfaces, Ceramic-on-metal and Metal-on-metal as Used in Cementless Primary Hip Arthroplasty
Brief Title: A Study Comparing Ceramic-on-metal Articulation to Metal-on-metal Articulation in Cementless Primary Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMETEU.CR.EU11
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Metal-on-Metal Joint Prostheses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceramic On Metal (Experimental): This arm utilizes the ceramic on metal articulation using the M2a-38™ mm cup.
  Interventions: Device: Ceramic On Metal
- Metal on Metal (Active Comparator): This arm utilizes the metal on metal articulation using M2a-38™ mm cup.
  Interventions: Device: Metal on Metal

INTERVENTIONS:
Device: Ceramic On Metal — Ceramic on Metal articulation using M2a-38™ mm cup
  Arms: Ceramic On Metal
Device: Metal on Metal — Metal on Metal articulation using M2a-38™ mm cup
  Arms: Metal on Metal

SUMMARY:
The aim of this study is to demonstrate the non-inferiority of the ceramic on metal articulation using M2a-38™ mm cup compared to the metal on metal articulation using the same cup.

DETAILED DESCRIPTION:
The aim of this study is to demonstrate the non-inferiority of the ceramic on metal articulation using M2a-38™ mm cup compared to the metal on metal articulation using the same cup in regards to the composite clinical success (CCS) rate, as defined in the protocol, at 2 year postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with osteoarthritis and suitable for primary Total Hip Replacement
* Patients preoperative Harris Hip Score <= 70 points
* Patients aged over 18 and under 75
* Patients with limited co-morbidity - ASA I-III
* Patients with normal urea and electrolyte levels and creatinine levels
* Patients must be able to understand instructions and be willing to return for follow-up
* Patients willing to provide blood and urine samples for metal ion analysis at follow up

Exclusion Criteria:

* Patients preoperative Harris Hip Score > 70 points
* Previous prosthetic hip surgery
* Patients with significant co-morbidity - ASA IV - V
* Dementia and inability to understand and follow instructions
* Neurological conditions affecting movement
* Existing metal implant or fixation device
* Pregnancy
* Presence of symptomatic arthritis in other lower limb joints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2009-05; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. Stranks, FRCS, Principal Investigator — North Hampshire Hospital; M Pesola, Principal Investigator — Central Finland Central Hospital; H Kauppinen, Principal Investigator — Kymenlaakso Central Hospital Kotka Finland
Locations (3):
- Finland (2):
  - Central Finland Central Hospital, Jyväskylä
  - Kymenlaakso Central Hospital, Kotka
- North Hampshire Hospital, Basingstoke, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Higgins JE, Conn KS, Britton JM, Pesola M, Manninen M, Stranks GJ. Early Results of Our International, Multicenter, Multisurgeon, Double-Blinded, Prospective, Randomized, Controlled Trial Comparing Metal-on-Metal With Ceramic-on-Metal in Total Hip Arthroplasty. J Arthroplasty. 2020 Jan;35(1):193-197.e2. doi: 10.1016/j.arth.2019.08.002. Epub 2019 Aug 22. PMID 31540737

RESULTS

PARTICIPANT FLOW:
Groups:
- Ceramic On Metal: Patients that underwent total hip arthroplasty, who received a M2a-38mm cup and the Biolox delta 38 mm ceramic femoral head.
- Metal on Metal: Patients that underwent total hip arthroplasty, who received a M2a-38mm cup and the 38 mm cobalt chromium molybdenum (CoCrMo) modular femoral head.
Period: Overall Study
Arm/Group | Ceramic On Metal | Metal on Metal
Started | 111 | 102
Completed | 56 | 53
Not Completed | 55 | 49

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceramic On Metal | Metal on Metal | Total
Number analyzed (Participants) | 111 | 102 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] — Age (years) at date of surgery
  years | 65.2 (7) | 65.3 (7.2) | 65.2 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 78
  Male | 73 | 62 | 135
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Finland | 30 | 22 | 52
  United Kingdom | 81 | 80 | 161

OUTCOME MEASURES:

1. Primary Outcome: Composite Clinical Success (CCS) Rate as Defined in the Protocol
Description: CCS is defined as:
  a. Total Harris Hip Score > 80 points, and b. No acetabular or femoral revision or removal, and c. No pending acetabular or femoral revision or removal as defined in radiographic evaluation by: i. An acetabular radiographic assessment with all of the following:
  1. Migration < 4 mm, and
  2. Change in angle of inclination < 4o, and
  3. Absence of osteolysis, and ii. A femoral radiographic assessment with all of the following:
  1. Subsidence < 5 mm, and 2. Absence of osteolysis.
  The HHS including a series of questions answered by the patient and physical examinations recorded by a qualified health care professional covers four domains: pain (one item, 0-44 points), function and functional activities (seven items, 0-47 points), absence of deformity (one item, 0-4 points) and range of motion (one item, 0-5 points). To obtain a final score, the points are summed. The outcome score can be categorized as Excellent: 90-100; Good: 80-90; Fair: 70-80; Poor: < 70
Time Frame: 2 years post-operatively
Population: Due to a lack of radiographic evaluation data, the overall number of participants analyzed is smaller than the actual number enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Ceramic On Metal | Metal on Metal
Number analyzed (Participants) | 75 | 77
Participants | 59 | 63

2. Secondary Outcome: Oxford Hip Score
Description: The Oxford Hip Score (OHS) is a patient-reported outcome measure that was developed to specifically assess the patient's perspective of outcome following THA. The OHS consists of twelve questions covering function and pain associated with the hip. To calculate the total score, each response is scored from 0 (worst outcome) to 4 (best outcome) and the sum of all 12 items is reported with a maximum of 48, representing the best score possible. The outcome score can be categorized as Excellent: > 41; Good: 34 - 41; Fair: 27 - 33; Poor: < 27.
Time Frame: pre-operatively, 6 weeks post-operatively, 6 months post-operatively, 1, 2, 3, 4, 5 and 10 years post-operatively
Population: 2 patients were not included in analysis due to receiving a different articulation (not the study device). Other than that, the number of participants decreased over time due to several reasons, such as missing visits or lost to follow-up or withdrawn from the study for any reason.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ceramic On Metal | Metal on Metal
Number analyzed (Participants) | 108 | 102
units on a scale
  preoperative | 22.7 (6.9) | 22.1 (7.3)
  6 weeks postoperative: number analyzed (Participants) | 105 | 99
  6 weeks postoperative | 37.3 (6.8) | 39.0 (6.7)
  6 months postoperative: number analyzed (Participants) | 104 | 99
  6 months postoperative | 45.0 (4.3) | 44.8 (5.2)
  1 year postoperative: number analyzed (Participants) | 104 | 98
  1 year postoperative | 46.0 (3.8) | 46.1 (4.1)
  2 years postoperative: number analyzed (Participants) | 99 | 91
  2 years postoperative | 46.6 (2.7) | 45.9 (4.5)
  3 years postoperative: number analyzed (Participants) | 71 | 71
  3 years postoperative | 46.4 (3.5) | 45.9 (4.5)
  4 years postoperative: number analyzed (Participants) | 51 | 60
  4 years postoperative | 46.8 (2.7) | 46.0 (4.2)
  5 years postoperative: number analyzed (Participants) | 87 | 83
  5 years postoperative | 46.1 (3.1) | 45.9 (3.8)
  10 years postoperative: number analyzed (Participants) | 54 | 50
  10 years postoperative | 44.0 (7.9) | 42.1 (10.2)

3. Secondary Outcome: Womac Score
Description: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC score) is a standardised patient reported outcome measure consisting of 24 items divided into 3 sub-sections: Pain (5 items), stiffness (2 items) and physical function or "Activities of Daily Living; ADL" (17 items). A higher score indicates a worse clinical outcome. The maximum score for each subsection is Pain: 20 - 0; Stiffness: 8 - 0; ADL: 68 - 0.
Time Frame: pre-operatively, 6 weeks post-operatively, 6 months post-operatively, 1, 2, 3, 4, 5 and 10 years post-operatively
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Ceramic On Metal | Metal on Metal
Number analyzed (Participants) | 108 | 102
Units on a scale
  Pain pre-operatively | 10.5 (3.3) | 11.5 (2.9)
  Pain 6 weeks post-operatively: number analyzed (Participants) | 106 | 99
  Pain 6 weeks post-operatively | 2.9 (3.0) | 2.4 (2.8)
  Pain 6 months post-operatively: number analyzed (Participants) | 104 | 99
  Pain 6 months post-operatively | 0.8 (1.9) | 0.7 (1.8)
  Pain 1 year post-operatively: number analyzed (Participants) | 104 | 98
  Pain 1 year post-operatively | 0.5 (1.4) | 0.3 (1.0)
  Pain 2 year post-operatively: number analyzed (Participants) | 99 | 91
  Pain 2 year post-operatively | 0.3 (1.2) | 0.5 (1.7)
  Pain 3 year post-operatively: number analyzed (Participants) | 71 | 70
  Pain 3 year post-operatively | 0.4 (1.1) | 0.5 (1.6)
  Pain 4 year post-operatively: number analyzed (Participants) | 52 | 61
  Pain 4 year post-operatively | 0.3 (1.1) | 0.6 (2.0)
  Pain 5 year post-operatively: number analyzed (Participants) | 86 | 83
  Pain 5 year post-operatively | 0.6 (1.6) | 0.7 (1.8)
  Pain 10 year post-operatively: number analyzed (Participants) | 56 | 50
  Pain 10 year post-operatively | 0.6 (1.9) | 0.6 (1.9)
  Stiffness pre-operatively | 4.0 (1.3) | 4.1 (1.5)
  Stiffness 6 weeks post-operatively: number analyzed (Participants) | 106 | 99
  Stiffness 6 weeks post-operatively | 1.9 (1.3) | 1.8 (1.3)
  Stiffness 6 months post-operatively: number analyzed (Participants) | 103 | 99
  Stiffness 6 months post-operatively | 0.6 (1.0) | 0.7 (1.2)
  Stiffness 1 year post-operatively: number analyzed (Participants) | 103 | 98
  Stiffness 1 year post-operatively | 0.4 (0.8) | 0.4 (0.9)
  Stiffness 2 year post-operatively: number analyzed (Participants) | 99 | 91
  Stiffness 2 year post-operatively | 0.2 (0.6) | 0.4 (0.9)
  Stiffness 3 year post-operatively: number analyzed (Participants) | 71 | 70
  Stiffness 3 year post-operatively | 0.3 (0.9) | 0.1 (0.6)
  Stiffness 4 year post-operatively: number analyzed (Participants) | 52 | 61
  Stiffness 4 year post-operatively | 0.2 (0.6) | 0.4 (1.1)
  Stiffness 5 year post-operatively: number analyzed (Participants) | 86 | 83
  Stiffness 5 year post-operatively | 0.7 (1.2) | 0.7 (1.3)
  Stiffness 10 year post-operatively: number analyzed (Participants) | 56 | 52
  Stiffness 10 year post-operatively | 0.7 (1.2) | 0.9 (1.4)
  ADL pre-operatively: number analyzed (Participants) | 107 | 100
  ADL pre-operatively | 32.1 (10.6) | 33.7 (9.3)
  ADL 6 weeks post-operatively: number analyzed (Participants) | 105 | 98
  ADL 6 weeks post-operatively | 12.6 (9.4) | 11.1 (10.0)
  ADL 6 months post-operatively: number analyzed (Participants) | 102 | 98
  ADL 6 months post-operatively | 3.8 (5.4) | 5.0 (7.7)
  ADL 1 year post-operatively: number analyzed (Participants) | 103 | 98
  ADL 1 year post-operatively | 3.2 (7.9) | 3.8 (6.8)
  ADL 2 year post-operatively: number analyzed (Participants) | 99 | 89
  ADL 2 year post-operatively | 2.7 (5.9) | 3.4 (6.6)
  ADL 3 year post-operatively: number analyzed (Participants) | 71 | 70
  ADL 3 year post-operatively | 2.9 (6.8) | 2.7 (5.9)
  ADL 4 year post-operatively: number analyzed (Participants) | 52 | 61
  ADL 4 year post-operatively | 2.5 (5.1) | 2.7 (5.5)
  ADL 5 year post-operatively: number analyzed (Participants) | 86 | 83
  ADL 5 year post-operatively | 3.5 (5.8) | 4.3 (7.6)
  ADL 10 year post-operatively: number analyzed (Participants) | 54 | 50
  ADL 10 year post-operatively | 5.1 (7.6) | 5.6 (8.8)

4. Secondary Outcome: Metal Ion Concentrations in Blood
Description: Chromium and Cobalt concentrations in blood are measured in measurement unit nmol/L. The change from baseline analysis is presented.
Time Frame: 6 months post-operatively, 1, 2, 3 and 5 years post-operatively
Population: Metal Ion analysis is only performed on a subset of the patients. Other than that, the number of participants fluctuates over time due to several reasons, such as missing visits or lost to follow-up or withdrawn from the study for any reason.
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | Ceramic On Metal | Metal on Metal
Number analyzed (Participants) | 38 | 35
nmol/l
  Chromium 6 months: number analyzed (Participants) | 36 | 34
  Chromium 6 months | -1.8 (16.9) | 1.9 (15.3)
  Chromium 1 year | 1.5 (25.4) | 17.5 (32.5)
  Chromium 2 years: number analyzed (Participants) | 30 | 34
  Chromium 2 years | 1.4 (13.9) | 18.8 (29.9)
  Chromium 3 years: number analyzed (Participants) | 18 | 17
  Chromium 3 years | -15.3 (7.3) | -13.4 (8.2)
  Chromium 5 years: number analyzed (Participants) | 31 | 31
  Chromium 5 years | 8.9 (29.3) | 19.1 (30.7)
  Cobalt 6 months: number analyzed (Participants) | 36 | 34
  Cobalt 6 months | 8.8 (8.7) | 26.8 (25.1)
  Cobalt 1 year | 16.3 (28.3) | 41.4 (77.8)
  Cobalt 2 years: number analyzed (Participants) | 30 | 34
  Cobalt 2 years | 12.3 (18.2) | 45.1 (45.5)
  Cobalt 3 years: number analyzed (Participants) | 21 | 20
  Cobalt 3 years | 13.0 (19.6) | 57.5 (61.4)
  Cobalt 5 years: number analyzed (Participants) | 31 | 31
  Cobalt 5 years | 17.7 (46.4) | 64.9 (64.0)

5. Secondary Outcome: Survivorship
Description: Survival of the implant based on the removal or intended removal of the device. The percentage of patients that still have the implant 10 years post-operative is presented here.
Time Frame: 10 years post-op
Measure: Count of Participants; unit: Participants
Arm/Group | Ceramic On Metal | Metal on Metal
Number analyzed (Participants) | 111 | 102
Participants | 99 | 88

ADVERSE EVENTS:
Time Frame: From surgery until the last study visit at 10 years post-op.
Description: ISO definitions are applicable. 211 operative cases (110 COM and 101 MOM) were available for the analysis.
Arm/Group | Ceramic On Metal | Metal on Metal
All-Cause Mortality (participants affected / at risk) | 16/110 | 13/101
Serious Adverse Events (participants affected / at risk) | 35/110 | 38/101
Other Adverse Events (participants affected / at risk) | 0/110 | 0/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceramic On Metal (N=110) | Metal on Metal (N=101)
Revision (Surgical and medical procedures) | 12 (12) | 14 (14) — One or more components revised
Cancer (General disorders) | 6 (7) | 5 (5)
Cardiovascular problems (Cardiac disorders) | 4 (4) | 5 (5)
Muculoskeletal problems (Musculoskeletal and connective tissue disorders) | 13 (13) | 11 (11)
Other (General disorders) | 5 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-09-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT00754520/Prot_SAP_000.pdf